CLINICAL TRIAL: NCT03620773
Title: IMPROVE-T2D Study: Impact of Metabolic Surgery on Pancreatic, Renal and Cardiovascular Health in Youth With Type 2 Diabetes
Brief Title: Impact of Metabolic Surgery on Pancreatic, Renal and Cardiovascular Health in Youth With Type 2 Diabetes
Acronym: IMPROVE-T2D
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0704
Record Dates: First submitted 2018-08-01; First posted 2018-08-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Bariatric Surgery Candidate; Nephropathy; Diabetic Kidney Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes Complications; Weight Loss; Diabetic Nephropathies; Adolescent Obesity; Pediatric Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Kidney Diseases; Diabetic Nephropathies; Diabetes Mellitus; Diabetes Complications; Weight Loss; Pediatric Obesity | interventions — p-Aminohippuric Acid; Iohexol; Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: All participants in this study will receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clinical Investigation (Other): Participants will include youth who are scheduled for, and will undergo, vertical sleeve gastrectomy (VSG) surgery at the Bariatric Surgery Clinic at Children's Hospital of Colorado.
  To understand how bariatric surgery affects renal function, all participants will undergo assessment of Glomerular Filtration Rate, (Iohexol Inj 300 mg/mL) and Effective Renal Plasma Flow (Aminohippurate Sodium Inj 20%). In addition, participants will undergo imaging assessment that includes renal Blood Oxygen Level Dependent (BOLD) and Arterial Spin Labeling (ASL) MRI.
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 mg/mL; Procedure: Vertical Sleeve Gastrectomy; Procedure: Renal Biopsy

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure effective renal plasma flow (ERPF)
  Other Names: Aminohippuric acid; Para-aminohippurate; Sodium 4-amino hippurate (PAH) inj 20% 2g/10 mL
Drug: Iohexol Inj 300 mg/mL — Diagnostic aid/agent used to measure glomerular filtration rate (GFR)
  Other Names: omnipaque 300
Procedure: Vertical Sleeve Gastrectomy — Participants will undergo vertical sleeve gastrectomy surgery, a laparoscopic bariatric surgery procedure designed for weight loss in obese patients
  Other Names: Bariatric Surgery
Procedure: Renal Biopsy — Minimally invasive outpatient procedure in interventional radiology to obtain renal tissue cores.
  Other Names: Kidney Biopsy

SUMMARY:
Type 2 diabetes (T2D) in youth is increasing in prevalence in parallel with the obesity epidemic. In the US, almost half of patients with renal failure have DKD, and ≥80% have T2D. Compared to adult-onset T2D, youth with T2D have a more aggressive phenotype with greater insulin resistance (IR), more rapid β-cell decline and higher prevalence of diabetic kidney disease (DKD), arguing for separate and dedicated studies in youth-onset T2D. Early DKD is characterized by changes in intrarenal hemodynamic function, including increased renal plasma flow (RPF) and glomerular pressure with resultant hyperfiltration, is common in Y-T2D, and predicts progressive DKD. Studies evaluating the two currently approved medications for treating T2D in youth (metformin and insulin) have shown these medications are not able to improve β-cell function over time in the youth. However, recent evidence suggests that bariatric surgery in adults is associated with improvements in diabetes outcomes, and even T2D remission in many patients. Limited data in youth also supports the benefits of bariatric surgery, regarding weight loss, glycemic control in T2D, and cardio-renal health. While weight loss is important, the acute effect of bariatric surgery on factors such as insulin resistance likely includes weight loss-independent mechanisms. A better understanding of the effects of bariatric surgery on pancreatic function, intrarenal hemodynamics, renal O2 and cardiovascular function in youth with obesity with or without diabetes is critical to help define mechanisms of surgical benefits, to help identify potential novel future non-surgical approaches to prevent pancreatic failure, DKD and cardiovascular disease.

The investigators' overarching hypotheses are that: 1) Y-T2D is associated with IR, pancreatic dysfunction, intrarenal hemodynamic dysfunction, elevated renal O2 consumption and cardiovascular dysfunction which improve with bariatric surgery, 2) The early effect of bariatric surgery on intrarenal hemodynamics is mediated by improvement in IR and weight loss, 3) Some aspects of cardio-renal-metabolic complications of T2D are related to obesity and others to T2D independent of obesity. To address these hypotheses, the investigators will measure GFR, RPF, glomerular pressure and renal O2, in addition to aortic stiffness, β-cell function and insulin sensitivity in youth ages 12-21 with T2D (n=40) and in (n=up to 10) youth with similar BMI but without diabetes, before and after vertical sleeve gastrectomy (VSG). To further investigate the mechanisms of renal damage in youth with T2D, two optional procedures are included in the study prior to vertical sleeve gastrectomy: 1) kidney biopsy procedure and 2) induction of induced pluripotent stem cells (iPSCs) to assess morphometrics and genetic expression of renal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Obese youth with and without T2D (≥50 kg) scheduled for VSG
* Weight <550 lbs.
* BMI ≥ 35 kg/m2
* Age 12-21 years
* HbA1c ≤ 12% for participants with T2D, HbA1c < 6.5% for participants with obesity

Exclusion Criteria:

* Obesity or T2D onset (diagnosis) > 18 years of age
* Prepubertal
* Anemia
* For participants undergoing the optional Parts 2-4 of visits 2 and 4, seafood or iodine allergy
* Pregnancy or breastfeeding
* Claustrophobia, implantable devices (MRI contraindications)
* Recent diabetic ketoacidosis or hyperosmolar hyperglycemia
* Other causes of diabetes other than T2D
* For participants undergoing the optional Parts 2-4 of visits 2 and 4, diuretics, sodium-glucose co-transport (SGLT) 2 or 1 blockers, daily NSAIDs or aspirin, sulfonamides, procaine, thiazolsulfone or probenecid, atypical antipsychotics or regular use of oral steroids

Additional exclusion criteria for participants undergoing Visit 4 part 4, the optional kidney biopsy:

* Evidence of bleeding disorder or complications from bleeding
* Use of aspirin, NSAIDS or other blood thinner that cannot be safely stopped for a sufficient time period before and after the biopsy so as to add no additional risk of bleeding
* Blood urea nitrogen (BUN) > 80 gm/dL
* INR > 1.4
* PTT > 35 seconds
* Hemoglobin (Hgb) < 10 mg/dL
* Platelet count < 100,000 / µL
* Uncontrolled or difficult to control hypertension (> 150/90 mmHg at the day of biopsy)
* eGFR < 40 mL/min/1.73m2
* Single kidney (either by history, documented by prior imaging or ultrasound performed prior to the biopsy)
* > 2 cm discrepancy between left and right kidney sizes based on largest longitudinal diameter determined by ultrasound performed prior to the biopsy.
* Kidney size: One or both kidneys < 9 cm
* Hydronephrosis or other important renal ultrasound findings such as significant stone disease
* Any evidence of a current urinary tract infection as indicated on day of biopsy
* Clinical evidence of non-diabetic renal disease
* Positive urine pregnancy test or pregnancy

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Pancreatic β-cell function | 4 hours (MMTT)
  Measured by Mixed Meal Tolerance Test (MMTT)
Pancreatic β-cell function | 4 hours (hyperglycemic clamp)
  Measured by blood draws during/after hyperglycemic clamp
Effective Renal Plasma Flow (ERPF) | 4 hours
  Measured by PAH clearance
Glomerular Filtration Rate (GFR) | 4 hours
  Measured by iohexol clearance

SECONDARY OUTCOMES:
Renal Perfusion | 10 min
  Measured by Arterial Spin Labeling (ASL) MRI
Renal Oxygenation | 60 min
  Measured by Blood Oxygen Level Dependent (BOLD) MRI
Aortic Stiffness & Wall Shear Stress | 30 min
  Measured by Aortic MRI

OTHER OUTCOMES:
Podocyte numerical density and number per glomerulus | 4 hours
  Measured by light microscopy from tissue obtained by renal biopsy
Foot process width of glomeruli | 4 hours
  Measured from tissue obtained by renal biopsy
Detachment and endothelial fenestration of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Podocyte volume of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Number and identity of RNA in kidney cells | 4 hours
  Measured from tissue obtained by renal biopsy
Epigenetic profiling | 4 hours
  Measured from tissue obtained by renal biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Petter Bjornstad, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided